CLINICAL TRIAL: NCT02369393
Title: Treatment of Depression: Efficacy and Efficiency of Two Self-administered Online Intervention Protocols Based on Behavioral Activation and Physical Activity
Brief Title: Efficacy of Two Internet Delivered Intervention Programs for Depression: Behavioral Activation vs Physical Activity
Acronym: PROMETEOII
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Jaume I (Other)
Collaborators: University of Valencia (Other); Universitat Politècnica de València (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UJaimeI06
Record Dates: First submitted 2015-02-16; First posted 2015-02-23 (Estimated); Last update posted 2023-07-11 (Actual); Status verified 2023-07

CONDITIONS: Major Depressive Disorder
Keywords: Internet based treatment; Depression; Efficacy; Cost-effectiveness; Behavioral Activation; Self-applied; Ecological Momentary Assessment; Physical Activity
MeSH Terms: conditions — Depressive Disorder, Major; Depression; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Behavioral Activation (Experimental): BA treatment for depression is a simple, cost-effective method. There is evidence that the behavioral component may be the active mechanism of change in cognitive-behavioral treatments of clinical depression. One of the main objectives of the treatment is to systematically increase exposure to positive activities, and thereby improve affect and corresponding cognitions. Treatment will be delivered through an Internet based treatment platform with mobile phone components (either integrated in the treatment platform or as a separate system). The core components are: 1) psycho-education, 2) identifying important values and significant activities, 3) activity structuring and scheduling, 4) relapse prevention. These will be delivered over 4 modules. There will be a minimal therapist support.
  Interventions: Behavioral: Behavioral Activation
- Waiting list control group (No Intervention): In the waiting list control group (WL), subjects will receive no treatment during 8 weeks. We will not interfere but we will monitor carefully through self-report. Then participants will be randomised to the two treatment groups.
- Physical Activity (Experimental): There is evidence to suggest that the addition of cognitive behavioral therapies, specifically exercise, can improve treatment outcomes for many patients. Exercise is a behavioral intervention that has shown great promise in alleviating symptoms of depression. The treatment will be delivered through an Internet based treatment platform with mobile phone components (either integrated in the treatment platform or as a separate system). The core components of the PA treatment are: 1) psychoeducation: understand the mental health benefits of physical activity, 2) learn about the types and amounts of physical activity recommended, 3) motivation to perform and maintain physical activities, 4) relapse prevention. These will be delivered over 4 modules. There will be a minimal therapist support.
  Interventions: Behavioral: Physical Activity

INTERVENTIONS:
Behavioral: Behavioral Activation — Behavioral Activation intervention promotes the involvement in meaningful activities close to personal values.
  Arms: Behavioral Activation
Behavioral: Physical Activity — Physical Activity intervention promotes the gradual increase of the frequency and intensity of PA levels, with special attention to motivational strategies.
  Arms: Physical Activity

SUMMARY:
To compare the clinical and cost-effectiveness of Behavioral Activation (BA) and Physical Activity (PA) for adults with major depressive disorder (MDD) or adjustment disorder with depressive symptomatology with a wait list control group (WL) in Spanish population.

DETAILED DESCRIPTION:
Research shows that in 2030 (Mathers and Loncar, 2006) depression will become one of the three leading causes of disability. Depression is a common mental disorder with a negative impact on mental well-being, quality of life, and social and work-related functioning both in the short and longer term.

Additionally, depression is associated with increased morbidity, mortality, health care utilization and health care costs. On a population level, depression is one of the most costly diseases. The economic costs of depression were estimated at €136.3 billion (EU25) in 2010 in the EU and are still rising. European health care systems face the challenge of improving access to cost-effective treatments while simultaneously working to sustain budgetary stability in times of economic austerity.

Internet-based depression treatment appears a very promising alternative to current routine depression treatment strategies. Meta-analyses have demonstrated the clinical effectiveness and potential cost-effectiveness of Internet-based treatment for depression in controlled research setting. Internet-based treatment thus has the potential to keep depression treatment affordable, as it enables mental health care providers to reach out to large populations needing depression treatment at a better cost-effectiveness, but with similar levels of clinical efficacy and quality of care.

In Spain the trial will be carried out in a community sample, comparing the clinical and cost-effectiveness of BA or PA with WL for adults with major depressive disorder (MDD) and adjustment disorder with depressive symptomatology. Respondents will be followed until 6 months after baseline (measures will be taken at BL, 3 months, and 6 months).

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years of age or older
* Meet DSM-IV diagnostic criteria for MDD and adjustment disorder confirmed by MINI International Neuropsychiatric Interview version 5.0 and SCID I
* A score of 5 or higher on the PHQ-9 screening questionnaire.

Exclusion Criteria:

* Current high risk for suicide according to the MINI Interview section C
* Serious psychiatric co-morbidity: substance dependence, bipolar affective disorder, psychotic illness, obsessive compulsive disorder, as established at the MINI interview
* Currently receiving psychological treatment for depression in primary or specialised mental health care
* Being unable to comprehend the spoken and written language (Spanish)
* Not having access to a PC and fast Internet connection (i.e. broadband or comparable).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2021-11-02 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Change in Patient Health Questionnaire-9 | Change from baseline to 2 months, 5 months, and 8 months
Change in the Beck Depression Inventory | Change from baseline to 2 months, 5 months, and 8 months

SECONDARY OUTCOMES:
Change in the EQ-5D-5L (EuroQol) | Change from baseline to 2 months, 5 months, and 8 months
Change in the Quality of Life (QLI) | Change from baseline to 2 months, 5 months, and 8 months
Change in the Overall Anxiety Severity and Impairment Scale (OASIS) | Change from baseline to 2 months, 5 months, and 8 months
Change in the Positive and Negative Affect Scale (PANAS) | Change from baseline to 2 months, 5 months, and 8 months
Change in the Happiness Scale (Fordyce) | Change from baseline to 2 months, 5 months, and 8 months
Change in the Satisfaction with Life Scale (SWLS, Diener) | Change from baseline to 2 months, 5 months, and 8 months
Change in the Ryff Scale of Psychological Wellbeing | Change from baseline to 2 months, 5 months, and 8 months
Change in the Behavioral Activation for Depression Scale - Short Form (BADS-SF) | Change from baseline to 2 months, 5 months, and 8 months
Change in the Environmental Reward Observation Scale (EROS) | Change from baseline to 2 months, 5 months, and 8 months
Change in Beck Depression Inventory (BDI-II) | Change from baseline to 2 months, 5 months, and 8 months

OTHER OUTCOMES:
Eysenck Personality Questionnaire-Revised Short Form (Neuroticism subscale) | Baseline
Credibility and expectancy questionnaire (CEQ) | 2 weeks
Self concordance motivation (SCM) | 2 weeks
Working Alliance Inventory (WAI-SF) | 3 weeks
System usability scale (SUS) | 2 months
Change in preferences for treatment scale (self-applied vs face to face) | Change from baseline to 2 months
Satisfaction with the treatment | 2 months
Change in the MINI International Neuropsychiatric Interview (M.I.N.I) version 5.0 | Change from baseline to 2 months
Change in Structured Clinical Interview (SCID-I) for Adjustment Disorders | Change from baseline to 2 months
Attitudes towards Psychological Online Interventions Questionnaire (APOI) | Baseline
Semi-structured interview about users´ intervention experience | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Botella, PhD, Principal Investigator — Universitat Jaume I;CIBERObn ISC III, Spain; Rosa Baños, PhD, Principal Investigator — Universitat de Valencia; CIBERObn ISC III, Spain
Locations (1):
- University Jaume I, Castellon, Spain

REFERENCES:
- [Background] Andersson G, Cuijpers P. Internet-based and other computerized psychological treatments for adult depression: a meta-analysis. Cogn Behav Ther. 2009;38(4):196-205. doi: 10.1080/16506070903318960. PMID 20183695
- [Background] Cavanagh K, Shapiro DA. Computer treatment for common mental health problems. J Clin Psychol. 2004 Mar;60(3):239-51. doi: 10.1002/jclp.10261. PMID 14981789
- [Background] Coffman SJ, Martell CR, Dimidjian S, Gallop R, Hollon SD. Extreme nonresponse in cognitive therapy: can behavioral activation succeed where cognitive therapy fails? J Consult Clin Psychol. 2007 Aug;75(4):531-41. doi: 10.1037/0022-006X.75.4.531. PMID 17663608
- [Background] Davidson TM, Yuen EK, Felton JW, McCauley J, Gros KS, Ruggiero KJ. Feasibility assessment of a brief, web-based behavioral activation intervention for adolescents with depressed mood. Int J Psychiatry Med. 2014;48(1):69-82. doi: 10.2190/PM.48.1.f. PMID 25354927
- [Background] Sudak DM, Majeed MH, Youngman B. Behavioral activation: a strategy to enhance treatment response. J Psychiatr Pract. 2014 Jul;20(4):269-75. doi: 10.1097/01.pra.0000452563.05911.c9. PMID 25036582
- [Background] Cuijpers P, Donker T, van Straten A, Li J, Andersson G. Is guided self-help as effective as face-to-face psychotherapy for depression and anxiety disorders? A systematic review and meta-analysis of comparative outcome studies. Psychol Med. 2010 Dec;40(12):1943-57. doi: 10.1017/S0033291710000772. Epub 2010 Apr 21. PMID 20406528
- [Background] Soucy Chartier I, Provencher MD. Behavioural activation for depression: efficacy, effectiveness and dissemination. J Affect Disord. 2013 Mar 5;145(3):292-9. doi: 10.1016/j.jad.2012.07.023. Epub 2012 Aug 9. PMID 22884236
- [Background] Churchill R, Moore TH, Furukawa TA, Caldwell DM, Davies P, Jones H, Shinohara K, Imai H, Lewis G, Hunot V. 'Third wave' cognitive and behavioural therapies versus treatment as usual for depression. Cochrane Database Syst Rev. 2013 Oct 18;(10):CD008705. doi: 10.1002/14651858.CD008705.pub2. PMID 24142810
- [Background] Dimidjian S, Barrera M Jr, Martell C, Munoz RF, Lewinsohn PM. The origins and current status of behavioral activation treatments for depression. Annu Rev Clin Psychol. 2011;7:1-38. doi: 10.1146/annurev-clinpsy-032210-104535. PMID 21275642
- [Background] Dimidjian S, Hollon SD, Dobson KS, Schmaling KB, Kohlenberg RJ, Addis ME, Gallop R, McGlinchey JB, Markley DK, Gollan JK, Atkins DC, Dunner DL, Jacobson NS. Randomized trial of behavioral activation, cognitive therapy, and antidepressant medication in the acute treatment of adults with major depression. J Consult Clin Psychol. 2006 Aug;74(4):658-70. doi: 10.1037/0022-006X.74.4.658. PMID 16881773
- [Background] Fitzsimons CF, Baker G, Gray SR, Nimmo MA, Mutrie N; Scottish Physical Activity Research Collaboration (SPARColl). Does physical activity counselling enhance the effects of a pedometer-based intervention over the long-term: 12-month findings from the Walking for Wellbeing in the west study. BMC Public Health. 2012 Mar 19;12:206. doi: 10.1186/1471-2458-12-206. PMID 22429600
- [Background] Azevedo Da Silva M, Singh-Manoux A, Brunner EJ, Kaffashian S, Shipley MJ, Kivimaki M, Nabi H. Bidirectional association between physical activity and symptoms of anxiety and depression: the Whitehall II study. Eur J Epidemiol. 2012 Jul;27(7):537-46. doi: 10.1007/s10654-012-9692-8. Epub 2012 May 24. PMID 22623145
- [Background] Loprinzi PD, Mahoney S. Concurrent occurrence of multiple positive lifestyle behaviors and depression among adults in the United States. J Affect Disord. 2014 Aug;165:126-30. doi: 10.1016/j.jad.2014.04.073. Epub 2014 May 5. PMID 24882189
- [Background] Goodwin RD. Association between physical activity and mental disorders among adults in the United States. Prev Med. 2003 Jun;36(6):698-703. doi: 10.1016/s0091-7435(03)00042-2. PMID 12744913
- [Background] Harvey SB, Hotopf M, Overland S, Mykletun A. Physical activity and common mental disorders. Br J Psychiatry. 2010 Nov;197(5):357-64. doi: 10.1192/bjp.bp.109.075176. PMID 21037212
- [Background] Hollon SD, Ponniah K. A review of empirically supported psychological therapies for mood disorders in adults. Depress Anxiety. 2010 Oct;27(10):891-932. doi: 10.1002/da.20741. PMID 20830696
- [Background] Jancey JM, Lee AH, Howat PA, Clarke A, Wang K, Shilton T. The effectiveness of a physical activity intervention for seniors. Am J Health Promot. 2008 May-Jun;22(5):318-21. doi: 10.4278/ajhp.22.5.318. PMID 18517091
- [Background] Johansson R, Andersson G. Internet-based psychological treatments for depression. Expert Rev Neurother. 2012 Jul;12(7):861-9; quiz 870. doi: 10.1586/ern.12.63. PMID 22853793
- [Background] King AC, Friedman R, Marcus B, Castro C, Napolitano M, Ahn D, Baker L. Ongoing physical activity advice by humans versus computers: the Community Health Advice by Telephone (CHAT) trial. Health Psychol. 2007 Nov;26(6):718-27. doi: 10.1037/0278-6133.26.6.718. PMID 18020844
- [Background] Lejuez CW, Hopko DR, Acierno R, Daughters SB, Pagoto SL. Ten year revision of the brief behavioral activation treatment for depression: revised treatment manual. Behav Modif. 2011 Mar;35(2):111-61. doi: 10.1177/0145445510390929. PMID 21324944
- [Background] Mead GE, Morley W, Campbell P, Greig CA, McMurdo M, Lawlor DA. Exercise for depression. Cochrane Database Syst Rev. 2009 Jul 8;(3):CD004366. doi: 10.1002/14651858.CD004366.pub4. PMID 19588354
- [Background] Fjeldsoe BS, Marshall AL, Miller YD. Behavior change interventions delivered by mobile telephone short-message service. Am J Prev Med. 2009 Feb;36(2):165-73. doi: 10.1016/j.amepre.2008.09.040. PMID 19135907
- [Background] Mota-Pereira J, Silverio J, Carvalho S, Ribeiro JC, Fonte D, Ramos J. Moderate exercise improves depression parameters in treatment-resistant patients with major depressive disorder. J Psychiatr Res. 2011 Aug;45(8):1005-11. doi: 10.1016/j.jpsychires.2011.02.005. Epub 2011 Mar 5. PMID 21377690
- [Background] Pinninti NR, Madison H, Musser E, Rissmiller D. MINI International Neuropsychiatric Schedule: clinical utility and patient acceptance. Eur Psychiatry. 2003 Nov;18(7):361-4. doi: 10.1016/j.eurpsy.2003.03.004. PMID 14643565
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Konig HH, Born A, Gunther O, Matschinger H, Heinrich S, Riedel-Heller SG, Angermeyer MC, Roick C. Validity and responsiveness of the EQ-5D in assessing and valuing health status in patients with anxiety disorders. Health Qual Life Outcomes. 2010 May 5;8:47. doi: 10.1186/1477-7525-8-47. PMID 20444251
- [Background] Newman MG, Szkodny LE, Llera SJ, Przeworski A. A review of technology-assisted self-help and minimal contact therapies for anxiety and depression: is human contact necessary for therapeutic efficacy? Clin Psychol Rev. 2011 Feb;31(1):89-103. doi: 10.1016/j.cpr.2010.09.008. Epub 2010 Oct 14. PMID 21130939
- [Background] Plonczynski DJ. Measurement of motivation for exercise. Health Educ Res. 2000 Dec;15(6):695-705. doi: 10.1093/her/15.6.695. PMID 11142077
- [Background] Stanton R, Reaburn P. Exercise and the treatment of depression: a review of the exercise program variables. J Sci Med Sport. 2014 Mar;17(2):177-82. doi: 10.1016/j.jsams.2013.03.010. Epub 2013 Apr 18. PMID 23602562
- [Background] Mammen G, Faulkner G. Physical activity and the prevention of depression: a systematic review of prospective studies. Am J Prev Med. 2013 Nov;45(5):649-57. doi: 10.1016/j.amepre.2013.08.001. PMID 24139780